CLINICAL TRIAL: NCT05457998
Title: BioFINDER-Brown: Examination of Alzheimer's Disease Biomarkers
Status: Enrolling by invitation | Type: Observational
Sponsor: Butler Hospital (Other)
Collaborators: The Warren Alpert Foundation (Unknown); Brown University (Other); University of Rhode Island (Other); Hoffmann-La Roche (Industry); Eli Lilly and Company (Industry); GE Healthcare (Industry)
Responsible Party: Principal Investigator, Edward Huey, Director, Memory and Aging Program, Butler Hospital; Martin M. Zucker Professor of Psychiatry and Human Behavior, Associate Director for Clinical Research, Brown Center for Alzheimer's Disease Research Alpert Medical School of Brown University, Butler Hospital
Other Study IDs: 1745146
Record Dates: First submitted 2022-07-11; First posted 2022-07-14 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment; Dementia
Keywords: Early diagnosis; Biomarker; PET; MRI; β-amyloid; tau; Cognitive test
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Dementia; Disease; Pick Disease of the Brain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Main study population: Cognitively unimpaired individuals (50-80 y): Participants will be enrolled based on a predetermined ratio of Alzheimer's Disease plasma and PET biomarker risk levels (e.g., as P-tau217 and amyloid PET).
  FOLLOW-UP FOR 4 YEARS: Cognitive testing, blood draws and retinal imaging will be conducted at baseline and 12 months. Cognitive testing and blood draws will be conducted at 24 months and 36 months.
  MRI and amyloid PET scans will be performed at screening/baseline and 24 months. An additional amyloid PET scan will be performed at 48 months.
  Interventions: Diagnostic Test: Flutemetamol F18 Injection
- Sub-group 1: Optional Tau PET imaging sub-study: An optional tau PET imaging sub-study will be conducted in 70 subjects from the main study population who elect to participate.
  If enrolled in the optional tau PET imaging sub-study, participants will have three tau PET scans with [18F]RO-948: at baseline, 24 months, and 48 months.
  Interventions: Diagnostic Test: [18F]-RO6958948 Injection
- Sub-group 2: Optional Tau PET tracer comparison sub-study: An optional tau PET tracer comparison sub-study will be conducted in 30 subjects from the main study population who elect to participate.
  Tau PET scans with 2 tracers ([18F]RO-948 and [18F]MK-6240) will be performed at baseline and 24 months. An additional Tau PET scan with [18F]RO-948 will be performed at 48 months.
  Interventions: Diagnostic Test: [18F]-RO6958948 Injection; Diagnostic Test: [18F]-MK-6240 Injection

INTERVENTIONS:
Diagnostic Test: Flutemetamol F18 Injection — PET imaging of Abeta amyloid
  Other Names: Vizamyl
  Groups: Main study population: Cognitively unimpaired individuals (50-80 y)
Diagnostic Test: [18F]-RO6958948 Injection — PET imaging of Tau aggregates
  Groups: Sub-group 1: Optional Tau PET imaging sub-study; Sub-group 2: Optional Tau PET tracer comparison sub-study
Diagnostic Test: [18F]-MK-6240 Injection — PET imaging of Tau aggregates
  Groups: Sub-group 2: Optional Tau PET tracer comparison sub-study

SUMMARY:
This research study aims to examine biomarkers of Alzheimer's disease as early as possible which could potentially be a screening tool for the general population. This observational study will take place at the Memory and Aging Program at Butler Hospital. The study will enroll up to 200 cognitively healthy subjects aged 50 to 80 years with ongoing recruitment and enrollment for 2 years, and subject participation lasting approximately 4 years. Disclosure of AD risk assessments will be an optional procedure. Two PET imaging sub-studies will also be optional.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between the ages of 50 and 80 years old (inclusive)
* Score of 16 or above on the MoCA telephone
* Score of 27 or greater on the MMSE for individuals aged 50 to 64 years old or a score of 26 or greater for individuals aged 65 to 80 years old
* Participants in the 50-60 age range will additionally need to meet at least one of the following: (1) First degree family history of dementia with onset before age 75; (2) APOE e4 allele carrier; or (3) Prior elevated result on amyloid PET or amyloid CSF testing
* Conversationally fluent in English to the extent that an interpreter is not necessary for comprehension of the study information, procedures, and cognitive tests.
* If participants elect to participate in the optional disclosure procedure, they will be required to have an appropriate study partner who agrees to participate in the study and who is intellectually, visually, and auditory capable, and conversationally fluent in English to the extent that an interpreter is not necessary.
* Adequate visual and auditory acuity to allow neuropsychological testing.
* Participants must be willing and able to provide written informed consent.

Exclusion Criteria:

* Diagnosis of mild cognitive impairment or dementia
* History of significant brain injury or other known neurologic disease or insult, resulting in lasting cognitive sequelae that would confound the assessment and staging of potential neurodegenerative disease (e.g., Huntington's disease, Parkinson's disease, Parkinsonism due to multiple system atrophy (MSA), progressive supranuclear palsy (PSP), Shy Drager Syndrome (SDS) or other neuro-degenerative dementias, encephalitis or other brain infection, epilepsy or stroke with lasting impairment to cognitive function).
* Current serious or unstable systemic illness or organ failure that, in the PI's judgement, would make it difficult to participate in the study (e.g., such as terminal cancer, cardiovascular, hepatic, renal, gastroenterological, respiratory, endocrinologic, neurologic, psychiatric, immunologic, or hematologic disease or other conditions ). History of cancer is acceptable with at least one year in remission with a good prognosis.
* Individuals with clinically significant depression, bipolar disorder, anxiety, or suicidal ideations within the past year as defined by the most current version of the Diagnostic and Statistical Manual of Mental Disorders (DSM).
* A history of schizophrenia as defined by the most current version of the DSM.
* History within the past year of chronic alcohol or drug abuse/dependence as defined by the most current version of the DSM.
* Marijuana use is acceptable, but frequent users will be asked to abstain from use within 24 hours of any assessments.
* Refusing or unable to complete any study procedures.
* Currently enrolled in another study which involves clinical drug trial or other medical intervention.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will be conducted in up to 200 subjects between the ages of 50-80 who are cognitively unimpaired. Participants must also pass all inclusion/exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-06-14 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Rate of change in plasma biomarkers | Time zero equals the baseline visit. All subjects will subsequently attend follow-up visits every year for 4 years after baseline.
  Validate and assess longitudinal changes from baseline in plasma amyloid, phosphorylated tau (p-tau) and other fluid biomarkers (e.g., neurofilament light).
Rate of change in cerebral amyloid pathology | Time Frame: Time zero equals the baseline visit. All subjects will subsequently attend follow-up visits every year for 5 years after baseline.
  Longitudinal assessment of cerebral amyloidosis based on amyloid PET imaging.
Rate of change in Tau PET measures | Time zero equals the baseline visit. All subjects will subsequently attend follow-up visits every year for 4 years after baseline.
  Longitudinal assessment of cerebral tau accumulation based on tau PET imaging.

SECONDARY OUTCOMES:
Rate of cognitive decline as measured by traditional cognitive and behavioral assessments | Time zero equals the baseline visit. All subjects will subsequently attend follow-up visits every year for 4 years after baseline.
Rate of cognitive decline as measured by digital cognitive assessments | Time zero equals the baseline visit. All subjects will subsequently attend follow-up visits every year for 4 years after baseline.
Rate of change in retinal imaging metrics | Time zero equals the baseline visit. All subjects will subsequently attend follow-up visits every year for 4 years after baseline.
Rate of change in psychological wellness as measured by the Geriatric Depression Scale | Time zero equals the baseline visit. All subjects will subsequently attend follow-up visits every year for 4 years after baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Edward Huey, MD, Principal Investigator — Butler Hospital Memory and Aging Program
Locations (1):
- Butler Hospital Memory and Aging Program, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Undecided